CLINICAL TRIAL: NCT01498341
Title: Hypoparathyroidism, Autosomal Dominant Hypocalcaemia and Pseudohypoparathyroidism in Denmark - Epidemiology, Causes, Symptoms and Prognoses
Brief Title: Hypoparathyroidism in Denmark
Acronym: HypoPT
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-20110074
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2013-01

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Epidemiology; Prognosis; Symptoms
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Biospecimen Retention: None Retained — 2 designs: Case-finding; Case-control
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify the number of persons in Denmark with the diagnose hypoparathyroidism, autosomal dominant hypocalcaemia or pseudohypoparathyroidism. Also the investigators want to identify the causes and symptoms of these patients and their prognosis.

DETAILED DESCRIPTION:
Hypoparathyroidism (HypoPT) is a relatively rare disease, where the level of parathyroid hormone (parat hormone [PTH]) cannot maintain a physiologically sufficient concentration of plasma calcium (P-Ca). This may be due to neck surgery (most frequently), congenital HypoPT, auto-immune destruction of the parathyroid gland, peripheral resistance to PTH, pseudoHypoPT or magnesium deficiency, by which PTH cannot be released from parathyroid gland.

Low plasma levels of P-Ca are registered by the calcium-sensing-receptors (CaSR) located e.g. in the gld. Parathyroid cell membranes and in the renal tubules, by which the flow of PTH into plasma increases, with normalization of P-Ca and decreasing P-phosphate to follow. By lack of PTH the renal synthesis of 1,25-dihydroxycholecalciferol is dismissed, with decreased bone turnover as a consequence.

Congenital causes of HypoPT are very rare and seen either sporadic or hereditary. The hereditary forms are more frequent in some areas of the world: founder-effect and familial marriages. Autoimmune HypoPT caused by mutations in the AIRE gene results in lack of negative selection of the T-cells in thymus. Autosomal dominant hypocalcaemia is caused by gain-of-function mutations in the G-protein receptor CaRS in the main cells in the parathyroid gland and kidney tubules. PseudoHypoPT is due to resistance in the target organs, despite high concentrations of PTH. The symptoms are shown by Albrights's hereditary osteodystrophy, (AOH), (maternal allel). PseudopseudoHypoPT is characterized by AOH, but without the typical biochemical findings (paternal allel).

The clinical manifestations of HypoPT depend on whether it occurs acute or chronic. The affected systems are the neuromuscular, ectodermal, ocular, cardia and neuropsychiatric system and manifest by increased neuromuscular irritability including weakness, muscle cramps, paresthesias of the lips, tongue, fingers and feet, memory loss, cardiac arrhythmias and heart insufficient headaches, and uncontrollable cramping muscle movements of the wrists and feet (carpopedal spasms) and possibly dry and scaling skin. In severe cases there may be cataract. In children symptoms may include malformations of the teeth. Due to high blood phosphorous levels, intracranial calcifications (basal ganglia), renal stones, and renal failure may develop. Studies have shown that HypoPT patients have reduced quality of life compared to a control group; more often have anxiety, depression and feel somatic. Furthermore, they have more physical symptoms like fatigue, ache, pain in the extremists and heart complaints.

The level of PTH decreases during pregnancy, while the level of 1,25-dihydroxycholecalciferol almost double due to placental and increased renal expression of 1α-hydroxylase with increased intestinal calcium absorption to follow, This improves maters calcium homeostasis why pregnant women should be monitored closely to prevent complications for the fetus.

Standard therapy includes treatment with calcium and 1alfa-hydroxylated forms of vitamin D (e.g. calcitriol or alphacalcidol) in order to relieve the symptoms associated with hypocalcaemia.

Aim The aim of the project is to identify the number of people in Denmark with HypoPT incl. autosomal dominant hypocalcaemia and pseudohypoparathyroidism (case-finding-study), identify possible complications, especially the prevalence of kidney disease, cardiovascular disease, neuropsychiatric disease, fertility, hospitalization required hypo- or hypercalcaemia, overall number of hospitalizations and mortality (case-control study).

Design The study is primarily conducted as a case finding study where patients with possible hypoparathyroidism are identified through registry extracts with subsequent validation of the diagnose (case-status) by reviewing their medical charts. Secondary there are preformed a case-control-study and a clinical characterization of patients with idiopathic hypoparathyroidism.

Definition (verification) of hypoparathyroidism: A patient is considered to have verified HypoPT when a person in question has been diagnosed with hypoparathyroid hypocalcaemia witch has made it necessary to treat with drug from pharmaceutical group A11CC (vitamin D), whom the person in question has redeemed a prescription for at least 2 times.

Patient materials The participants are selected through two registry studies (search strategies) see flowcharts. The first register study is via the National Patient Register, while the second search is based on the Medicine Database.

Data extraction: For individuals identified through one of the two search strategies the following information are requested through the National Patient Registry, the Registry of Abortion, the Death Registry and the CPR Registry. All diagnose codes (from 1977-today), vital status, information about fertility and in case of death, the cause of death.

Data processing: All patients who have been identified though one of the above-mentioned data extraction will have copy of their journals, discharge summary and blood samples required concerning verification of the diagnose. In case of doubt the general practitioner can be contacted. For patients with a verified diagnose sex, birth data, time of onset and the cause of the disease will be registered. For patients with idiopathic HypoPT data about the examinations conducted to clarify the possible causes of the disease are also recorded.

To clarify the possible complications (comorbidity) to HypoPT, including the diseases influence on the patient's life expectancy a matched control population is requested from the CPR Registry. For each case with verified HypoPT 3 random control person matched on sex and age are withdrawn. For the control group a data extraction corresponding to the extraction on the patients with HypoPT are made. For both the patients with HypoPT and the control group the diagnoses are verified through review of journals and medical summaries. In case of doubt the general practitioner can be contacted. Besides clarifying the overall mortality and co-morbidity a stratified analysis of co-morbidity is conducted separated on ATC-groups with focusing on the cardiovascular, renal and neuropsychiatric complications. Stratification will also be conducted on reasons for developing HypoPT.

Research biobank The withdrawn blood samples will be stored in a research biobank for 15 years. The participants will be asked to give consent for this purpose. In addition they will be requested to give consent so the biological material can be used for further research upon specific approval by the local ethical committee. The biobank will be notified to the Danish Data Protection Agency under applicable law.

Statistic There will be calculated prevalence and incidence with corresponding 95 % confidence interval, CI, and mortality. Since the presence of HypoPT in Denmark and worldwide is unknown, it is not possible to perform power calculations for the case-control study.

ELIGIBILITY:
Inclusion Criteria for the case-control-study:

* Idiopathic hypoparathyroidism
* Pseudohypoparathyroidism
* Autosomal dominant hypocalcaemia

Exclusion Criteria for the case-control-study:

* Chronic kidney insufficience (creatinine above 200 umol/l)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population are persons with hypoparathyroidism, automalt dominant hypocalcaemia and pseudohypoparathyroidism.
  The population is selected via the National Danish Health Registre and the Danish Medical Registre
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Frequency of hypoparathyroidism, pseudohypoparathyroidism and autosomal dominant hypocalcaemia and its consequences | One year
  The frequency of hypoparathyroidism, pseudohypoparathyroidism and autosomal dominant hypocalcaemia. The frequence is estimated via the National Danish Health Register.
  The prevalence of kidney-, cardiovascular- and neuropsychiatric disease, fertility, hospitalization required hypo- or hypercalcaemia, overall number of hospitalizations and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, DmSci, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Internal Medicine and Endocrinology, Aarhus University Hospital, Tage-Hansens Gade, Aarhus, Region Midt, Denmark